CLINICAL TRIAL: NCT04928118
Title: Characterization Of The Hemodynamic Effects Of Impella On Renal Blood Flow And Oxygen Delivery And Risk Of Contrast-Associated Acute Kidney Injury Among Patients Undergoing Protected Percutaneous Coronary Intervention
Brief Title: Hemodynamic Effects Of Impella On Renal Circulation And Risk Of CA-AKI Among Patients Undergoing Protected PCI
Status: Withdrawn | Type: Observational
Why Stopped: PI may be leaving the institution
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HM20021800
Record Dates: First submitted 2021-05-26; First posted 2021-06-16 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Contrast-induced Acute Kidney Injury (CI-AKI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Impella protected Percutaneous coronary intervention (PCI): Patients undergoing Impella protected PCI as deemed necessary by interventional cardiologist - VCU Medical Center case based standard of care
  Interventions: Other: Evaluate the blood flow and pressure into kidneys

INTERVENTIONS:
Other: Evaluate the blood flow and pressure into kidneys — Renal artery pressure and flow measures will be obtained using dedicated equipment positioned into the renal artery under fluoroscopic guidance.
  A pulmonary artery catheter will be used to measure the pressure inside participant's renal vein and to collect small blood samples to measure oxygen content.

SUMMARY:
Patients undergoing Percutaneous Coronary Intervention (PCI) are exposed to the risk of suffering from a damage to the kidneys which goes under the name of Contrast-Associated Acute Kidney Injury (CA-AKI), which is more common if the subject has advanced heart or kidney disease. Up to 1 high risk patient in 3 can suffer from CA-AKI. Impella is a pump which sustain the heart in the course of PCI in high risk individuals. Incidentally, Impella was shown to also reduce the incidence of CA-AKI. The reason why Impella protects the kidneys is not currently known. The investigators aim at understanding it through measurements of kidney blood flow and metabolism.

DETAILED DESCRIPTION:
Contrast-associated acute kidney injury (CA-AKI) is among the major determinants of morbidity after percutaneous coronary intervention (PCI). Patients undergoing complex, high-risk indicated procedures (CHIP) are exposed to an increased risk of CA-AKI. Recent observational data suggested that mechanical circulatory support (MCS) with Impella in the course of CHIP PCI, i.e. Impella-protected PCI, may abate the risk of CA-AKI. A direct effect of MCS in improving renal perfusion has been postulated, but mechanistic evidence on the pathophysiologic effects of Impella on kidney hemodynamics is lacking. The investigators hypothesize that such improved renal outcomes during Impella protected PCI are attributable to increased blood flow as well as increased oxygen delivery to the kidneys granted by MCS. The aim of the present study is to fully characterize the renal hemodynamics as well as renal oxygen delivery and consumption during Impella-protected PCI using state-of-the-art invasive measurements, and to correlate those with functional magnetic resonance imaging of the kidney.

ELIGIBILITY:
Inclusion Criteria:

Impella-protected PCI selection criteria according to Virginia Commonwealth University (VCU) Complex PCI Program

* Left ventricular ejection fraction (LVEF) ≤35% and ≥1 complexity feature
* LVEF ≤45% and estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2 and ≥1 complexity feature
* LVEF ≤45% and eGFR 31-45 ml/min/1.73 m2 and ≥2 complexity features

Complexity features

* Planned treatment of ≥2 vessels
* Left main PCI
* Bifurcation intervention with 2-stent strategy
* Planned use of atherectomy (rotational, orbital, laser)
* Chronic total occlusion PCI
* PCI on last remaining vessel
* LVEDP >18 mmHg
* Cardiac index <2.0 l/min/m2 or pulmonary artery O2 saturation <55%

Exclusion Criteria:-

* Pregnancy or lactation
* Presence of non-MRI compatible implanted medical device
* Known absolute contraindication to Impella insertion, e.g. severe peripheral arterial disease, left ventricular thrombus, aortic mechanical prosthesis, or severe aortic valve stenosis
* Chronic hemodialysis before the index procedure
* Status post-renal transplant
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to undergo Impella assisted PCI procedure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Renal blood flow (RBF) | during PCI up to 5 hours
  thermodilution will be used to measure patterns of RBF in milliliters per minute

OTHER OUTCOMES:
Acute Kidney Injury (AKI) | up to 72 hours after PCI
  Change in creatine will be used to identify AKI
Anatomical changes | 3 days
  Pre and post-procedural kidney magnetic resonance imaging (MRI) will be used to explore any changes in acute renal ischemia due to the procedure
Renal oxygen delivery (ROD) | during PCI up to 5 hours
  ROD is defined as O2 content (CaO2) (RBF x CaO2). Blood samples during the procedure will be used to observe the patterns.
Renal oxygen consumption (ROC) | during PCI up to 5 hours
  ROC is defined as CaO2 and renal vein oxygen content (CvO2) as RBF x (CaO2 - CvO2). Blood samples during the procedure will be used to observe the patterns.
Renal oxygen extraction (ROE) | during PCI up to 5 hours
  ROE is defined as CaO2 and CvO2 as (CaO2 - CvO2)/CaO2. Blood samples during the procedure will be used to observe the patterns.
Renal vascular resistance (RVR) | during PCI up to 5 hours
  RVR will be calculated using mean arterial pressure (MAP) and renal vein pressure (RVP) as (MAP - RVP)/RBF.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Azzalini, MD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No